CLINICAL TRIAL: NCT04055857
Title: Structural and Functional Changes in Neuronal Intranuclear Inclusion Disease: A Pioneer Multi-modal 7T MRI Observational Study.
Brief Title: Structural and Functional Changes in Neuronal Intranuclear Inclusion Disease(NIID)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Collaborators: Zhejiang University Interdisciplinary Institute of Neuroscience and Technology (Unknown)
Responsible Party: Sponsor
Other Study IDs: 7TMRINIID
Record Dates: First submitted 2019-07-31; First posted 2019-08-14 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-06

CONDITIONS: Neuronal Intranuclear Inclusion Disease
MeSH Terms: conditions — Neuronal intranuclear inclusion disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NIID: NIID patients
- HC: healthy control

INTERVENTIONS:
Other:  — There is no Intervention.

SUMMARY:
To discover the microstructure, macrostructure and functional changes with 7T multi-modal magnetic resonance imaging of Neuronal Intranuclear Inclusion Disease, and to explore new biomarkers for evaluating the severity and the progression of Neuronal Intranuclear Inclusion Disease.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with NIID
2. Older than 18 years;
3. Sign the informed consent form.

Exclusion Criteria:

1. The informed consent is withdrawn by the subject;
2. Contraindications or intolerance to MRI: metallic foreign bodies, instability of vital signs, epilepsy, claustrophobia, etc.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects enrolled in the study shall be selected from NIID patients who are diagnosed with skin biopsy and gene detection. The Investigator is responsible for screening potential subjects and selecting those who meet the eligibility criteria for the study as described.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-07-31 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
fractional anisotropy (FA) | baseline
  Parameters to describe integrity of white matter in diffusion MR Imaging
mean diffusivity (MD) | baseline
  Parameters to describe integrity of white matter in diffusion MR Imaging
Intracellular volume fraction(icvf) | baseline
  Parameters to describe integrity of white matter in diffusion MR Imaging
orientation dispersion index (ODI) | baseline
  Parameters to describe integrity of white matter in diffusion MR Imaging
fiber number(fiber pass through the lesions) | baseline
  Parameters to describe integrity of white matter in diffusion MR Imaging
fractional anisotropy (FA) | 6 months
  Parameters to describe integrity of white matter in diffusion MR Imaging
mean diffusivity (MD) | 6 months
  Parameters to describe integrity of white matter in diffusion MR Imaging
Intracellular volume fraction(icvf) | 6 months
  Parameters to describe integrity of white matter in diffusion MR Imaging
orientation dispersion index (ODI) | 6 months
  Parameters to describe integrity of white matter in diffusion MR Imaging
fiber number(fiber pass through the lesions) | 6 months
  Parameters to describe integrity of white matter in diffusion MR Imaging
short-range and long-range functional connectivity around the lesions at rest | baseline
  Functional network connectivity impairments in patients
short-range and long-range functional connectivity around the lesions at rest | 6 months
  Functional network connectivity impairments in patients

CONTACTS AND LOCATIONS:
Overall Officials: Ruiliang Bai, Doctor, Principal Investigator — Zhejiang University Interdisciplinary Institute of Neuroscience and Technology (ZIINT); Hui Liang, Doctor, Principal Investigator — Zhejiang University
Locations (1):
- Siemens 7T MR, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No